CLINICAL TRIAL: NCT02261870
Title: "Detection of Acute Rejection in Heart Transplant Patients by Mean of T2 Quantification With MRI" Open Transversal Clinical Trial With Repeated Measures
Brief Title: Detection of Acute Graft Rejection in Heart Transplant Patients by Estimation of T2
Acronym: DRAGET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00848-39; CIC1433 (Other: 12-109_DRAGET)
Record Dates: First submitted 2014-09-25; First posted 2014-10-10 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Acute Graft Rejection; Heart Transplantation
Keywords: MRI, T2 quantification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALL_patients (Experimental): MRI T2 quantification : heart transplant patients will have 4-6 MRI exams for T2 quantification during their first year after transplantation.
  Interventions: Device: MRI T2 quantification

INTERVENTIONS:
Device: MRI T2 quantification — MRI acquisitions will be performed according to the already described method based on conventional Fast Spin Echo sequences and with an additional calibration pad positioned on the patient thorax (dedicated pad made by the Nancy CIC-IT with stable and adapted T2). MRI will be performed if possible before the biopsy and otherwise the radiologist will be kept blinded of the biopsy results.

SUMMARY:
The investigators propose a simple and non-invasive method to monitor heart transplant patients with MRI. Its diagnostic and prognostic values have already been assessed in two monocentric studies. Other monocentric studies based on related methods have confirmed the investigators findings. These studies are insufficient to allow a large diffusion of the technique. Only a large multi-centric study will change medical practices. In addition, this project will spread the new method at a national level and will allow an assessment of its practical usefulness in centres not familiar with MRI T2 quantification.

Furthermore, MRI seems to detect rejections at earlier stage than biopsy. A confirmation of this observation could lead to a modification of diagnostic criteria of cardiac graft rejection. The ultimate aim of the DRAGET project is to replace a strategy based solely on biopsy with one based on a first-line MRI (with biopsy only when needed) for a more efficient and earlier detection of rejection. This would constitute a major advance in patients security and comfort as well as an economic improvement.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patient
* Able to realize 4 couples Biopsy/MRI within 12 months after the transplant
* Mandatory enrolment in a social security plan
* Patient having signed an informed consent.

Exclusion Criteria:

* Contraindication to MRI: pacemaker, ferromagnetic foreign body, etc
* Impossibility to undergo MRI: claustrophobia, morbid obesity, hospitalisation in intensive care unit, arrhythmia
* Pregnancy
* Patients under a measure of legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of myocardial T2 assessed with MRI for the diagnosis of histological heart graft rejection (with 95% confidence interval). | 3 years after first inclusion
  endpoint = sensitivity and specificity acute rejection means presence of damaged myocytes in endomyocardial biopsy (former grade 2, grade 2R and grade 3R)

SECONDARY OUTCOMES:
Incidence of histological or clinical rejection within months of a couple MRI/biopsy with normal biopsy (grade<2R). | 3 years after first inclusion
  endpoint = number of rejections For this purpose, rejection will be defined as: a) acute rejection documented by presence of damaged myocytes in endomyocardial biopsy (former grade 2, grade 2R and grade 3R), or b) marked decrease in left ventricle ejection fraction (>10%), reversible after subsequent increase in immunosuppressive treatment.
Complications with MRI and with biopsies. | 3 years after first inclusion
  endpoint = Number of adverse events due to both exams
Magnitude of better tolerability of MRI over biopsies for the patient. | 3 years after first inclusion
  endpoint = Physical and psychological distress assessed by questionnaire using Likert scales. This questionnaire will be completed by the patients.
Inter-observer reproducibility of T2 quantification with MRI and of pathological grading of the biopsies. | 3 years after first inclusion
  endpoint = 95% interobserver limit of agreement for T2 quantification and Cohen's Kappa coefficient for histological grading.
Level of confidence, at the end of the study, of the expert-physicians of each centre concerning the use of T2 quantification as an alternative to routine biopsies. | 3 years after first inclusion
  endpoint = Confidence assessed by questionnaire using Likert scales. This questionnaire will be completed by study investigators at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Bonnemains, MD, PhD, Principal Investigator — INSERM, IADI U47, Nancy, France
Locations (10):
- France (10):
  - Hospices Civils de Lyon, Bron
  - CHU Grenoble, La Tronche
  - CHRU Nancy Brabois, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - CHU Bordeaux, Pessac
  - CHU de Rennes, Rennes
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - CHU de Tours, Tours

REFERENCES:
- [Derived] Bonnemains L, Cherifi A, Girerd N, Odille F, Felblinger J. Design of the DRAGET Study: a multicentre controlled diagnostic study to assess the detection of acute rejection in patients with heart transplant by means of T2 quantification with MRI in comparison to myocardial biopsies. BMJ Open. 2015 Oct 29;5(10):e008963. doi: 10.1136/bmjopen-2015-008963. PMID 26515686